CLINICAL TRIAL: NCT06225856
Title: An Open-Label, Multicenter, Phase I Study to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of YY201 in Patients With Advanced Solid Tumors and Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yuyao Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-YY201-CH1
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Tumor; Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study treatment (Experimental): Method of Administration: Single dose period: Single oral administration under fasting state; Multiple dose period: Oral administration under fasting state, QD.
  Interventions: Drug: YY201

INTERVENTIONS:
Drug: YY201 — Oral administration under fasting state.

SUMMARY:
This is a multicenter, open-label, phase I clinical study of YY201 in the patients with relapsed/refractory lymphomas and relapsed/refractory large granular lymphocytic leukemia who failed or cannot tolerate standard treatment.

DETAILED DESCRIPTION:
This study includes a dose escalation phase and a dose expansion phase. In the dose escalation phase the MTD and/or RP2D of YY201 will be determined and in the dose expansion phase the anti-tumor efficacy of YY201 will be evaluated in patients with relapsed⁄refractory hematological malignancies. The two-phase study will assess the preliminary anti-tumor efficacy , safety, tolerability, and PK profile of YY201 .

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients fully understand and sign ICF, voluntarily participate in the study, and able to follow and complete all study procedures.
* 2.Aged 18-80 years (including upper and lower limits), male or female.
* 3. The standard treatment failure (disease progression after treatment or treatment side effects not tolerance), or top treatment, or shall not apply to the current standard treatment for patients with:

  * Surgical excision is confirmed by histology or cytology can't or metastatic patients with advanced solid tumor;
  * Patients with relapsed or refractory hematologic malignancies
* 4. For patients with advanced solid tumors (dose-escalation phase), at least one tumor lesion that could be evaluated according to RECIST, version 1.1; (Dose-expansion phase) At least one measurable tumor lesion according to RECIST, version 1.1 (a tumor that is located in the previously irradiated area or another locoregional treatment site and is generally not considered a measurable lesion unless there is definite progression or persistence beyond 3 months of radiation).
* 5. In the dose-expansion phase, enrollment was limited to:

  * Advanced solid tumors (predominantly triple-negative breast cancer, pancreatic cancer, and head and neck squamous cell carcinoma) that are sensitive to STAT3 therapy;
  * Peripheral T-cell lymphoma (PTCL) with STAT3 mutation refractory to or relapsed after at least one or more lines of systemic therapy;
  * For patients with PTCL, computed tomography performed within 28 days before study entry should show at least one measurable tumor lesion in two vertical directions, with nodal lesions > 1.5cm in greatest dimension and extranodal lesions > 1.0cm (according to the 2014 lugano criteria).
  * Relapsed/refractory acute myeloid leukemia that is sensitive to STAT3 therapy, excluding acute promyelocytic leukemia (APL) and other secondary AML (e.g., MDS transformation, CML in blast phase, etc.)
* 6. ECOG physical condition≤1.
* 7. Patients with advanced primary liver cancer should meet the Child-Pugh liver function grading: grade A and better grade B (≤7).
* 8. Regular check need to meet the following requirements:

  * For advanced solid tumors, adequate bone marrow, liver, and kidney function is required:

    1. Blood system within 14 days (not received blood transfusions or hematopoietic stimulating factor treatment):

       Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥75×10^9/L; Hemoglobin (Hb) ≥85g/L;
    2. Liver function:

       Total bilirubin (TBIL) ≤1.5×ULN; Alanine aminotransferase (ALT) ≤3×ULN; Spread to the liver or liver cancer patient: 5 or less x ULN; Aspartate aminotransferase (AST) or less 3 x ULN; Spread to the liver or liver cancer patient: 5 or less x ULN;
    3. Renal function:

       Creatinine (Cr) or less 1.5 x ULN; Creatinine clearance (Ccr) (calculated only when creatinine > 1.5× ULN) ≥50ml/min (calculated according to Cockcroft-Gault formula, see Annex 2 of the protocol);
    4. Blood coagulation function:

       Activated partial thromboplastin time (APTT) ≤1.5×ULN; International normalized ratio (INR) ≤1.5×ULN;
    5. Urinary protein:

       Urine routine /24 hours urine protein qualitative ≤1+; Or urine protein qualitative ≥2+, 24 hours urine protein < 1g;
  * For patients with PTCL, routine blood hemoglobin or 80 g/L, neutrophils acuity 1.0 x 10^9 / L, 75 x 10^9 or higher platelet/L (within 14 days before test without blood transfusion or the use of biological stimulating factor);
  * For patients with AML, white blood cell counts ≤25 ×10^9/L (Hydroxyurea was allowed but not for 3 days before administration of the trial drug);
* 9. Agreed to provide archival tumor-tissue specimens or fresh tissue samples (Dose-expansion phase)
* 10.Expected survival of at least 3 months.
* 11. Women of childbearing potential had to have a negative serum or urine pregnancy test within 7 days before the first dose. Fertile male or female patients voluntarily during the study period and at the end of the study drug within 30 days of using effective birth control methods, such as abstinence, the double protective screen type cuts, condoms, contraceptive method of oral or injected contraceptives, intrauterine device, etc. All female patients will be considered fertile unless the female patient has undergone natural menopause, artificial menopause, or sterilization (e.g., hysterectomy, bilateral adnophorectomy, or radioactive ovarian irradiation).

Exclusion Criteria:

* 1. The adverse reactions of previous antineoplastic therapy have not recovered to CTCAE 5.0 grade ≤1 (except for toxicities without safety risks judged by investigators, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stable with hormone replacement therapy);
* 2. Clinically symptomatic parenchymal or leptomeningeal metastases that were judged by the investigator to be ineligible for enrollment and, for AML patients, known central nervous system (CNS) involvement
* 3. Within 4 weeks before delivery for the first time received chemotherapy, radiation therapy, biological therapy and endocrine therapy, immune therapy, such as antitumor drugs, with the exception of the following situations:

  * Nitrosourea or mitomycin C within 6 weeks before first use of study drug;
  * Oral fluorouracils and small-molecule targeted agents are administered 2 weeks before first use of the study drug or within the five half-lives of the drug, whichever is longer;
  * Have antitumor indications for the study of the first use of drugs of traditional Chinese medicines before 2 weeks;
  * For peripheral blood leukocyte count (WBC > 25 x 10^9 / L) of the patients, allowing use in treatment of the former and YY201 hydroxyurea control peripheral blood leukocytes;
  * Prophylactic intrathecal chemotherapy (cytarabine, dexamethasone, and methotrexate) unless it is used to prevent central leukemia.
* 4. Received other unlisted investigational drugs or treatments within 4 weeks before the first dose;
* 5. Previously received STAT3 inhibitor for anti-tumor treatment;
* 6. Major organ surgery (excluding needle biopsy) within 4 weeks before the first dose of medication or requiring elective surgery during the trial;
* 7. Uncontrolled malignant pleural, ascites, or pericardial effusion that was judged by the investigator to be ineligible for enrollment;
* 8.Unable to oral drug swallowing, or by the researchers determine the condition of the seriously affect the gastrointestinal tract absorption, including but not limited to, such as inflammatory bowel disease (crohn's disease and ulcerative colitis, for example), or malabsorption syndrome, or chronic diarrhea;
* 9. Patients who received a potent inducer or inhibitor of CYP3A4 within 1 week before the first dose or who required continued treatment with these drugs during the study;
* 10. Patients with active gastric and duodenal ulcer, ulcerative colitis and other gastrointestinal diseases, or unresected tumor with active bleeding, or other conditions that may cause gastrointestinal bleeding or perforation as judged by the investigator;
* 11. Thromboembolic events (including stroke events and/or transient ischemic attack) occurred within 12 months before the first dose of medication;
* 12. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months before the first dose of medication; Congestive heart failure with New York Heart Association (NYHA) grade ≥2; Left ventricular ejection fraction (LVEF) <50%; A history of primary cardiomyopathy, clinically significant prolongation of the QTc interval, or a screening QTc interval >470ms in women and >450ms in men;
* 13. Patients with active or previous autoimmune diseases with potential recurrence (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), excluding patients with clinically stable autoimmune thyroid diseases and type I diabetes mellitus;
* 14. Prior immunotherapy with grade ≥3 irAE or grade ≥2 immune-related myocarditis;
* 15. Researchers to determine the clinical significance of 3 or more electrolyte abnormalities
* 16. Patients with active infection requiring antiinfective treatment or unexplained fever (body temperature >38.5 ° C) during screening or before the first dose of medication;
* 17. Patients with active pulmonary tuberculosis (TB) who are receiving anti-TB treatment or have received anti-TB treatment within 1 year before the first dose; Known human immunodeficiency virus (HIV) infection; Patients with a history of hepatitis B were in the stage of active infection (HBsAg positive and HBV-DNA > the detection limit of the research center); Patients with a history of hepatitis C were in the active infection stage, defined as positive HCV antibody test and HCV RNA above the local detection cut-off value;
* 18. Patients who have received hematopoietic stem cell transplantation (HSCT) within 60 days prior to the start of study treatment, or are receiving immunosuppressive therapy after HSCT at screening, or have graft-versus-host disease (GVHD) requiring drug control:

  •Patients treated with fixed oral dose and/or topical corticosteroids for cutaneous GVHD may be enrolled with approval of the Sponsor.
* 19. Women who are pregnant (positive pregnancy test within 14 days before medication) or are breastfeeding.
* 20. Men with fertility needs;
* 21. Patients with known alcohol or drug dependence;
* 22. Patients judged by the investigator that may not be able to comply with all study procedures;
* 23. Any other disease, metabolic abnormality, abnormal physical examinations or laboratory abnormality with significant clinical significance. Investigator reasonably suspects that the patient has a disease or state that is not suitable for using of the study drug, or will affect interpretation of study results, or put the patient at high risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Up to 31 days after the initial drug administration
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0)
Maximum tolerated dose | Up to approximately 24 months
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of YY201 . The type, frequency and severity of TEAE will be evaluated during the treatment of YY201 .
Recommended Dose for Phase II Clinical Studies (RP2D) | Up to 31 days after the initial drug administration
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of YY201.

SECONDARY OUTCOMES:
Cmax | Up to 31 days after the initial drug administration
  Maximum serum concentration (Cmax) of YY201 will be investigated.
Tmax | Up to 31 days after the initial drug administration
  Time to maximum serum concentration (Tmax) of YY201 will be investigated.
T1/2 | Up to 31 days after the initial drug administration
  Half-life (T1/2) of YY201 will be investigated.
Duration of Response(DoR) | Up to approximately 24 months
  The time from the patient's first objective response to the patient's disease recurrence, progression, or death.
Time to Disease Response(TTR) | Up to approximately 24 months
  The time from the first dose of YY201 to the first occurrence of objective response.
Overall Survival (OS) | Up to approximately 24 months
  The time from start date of study drug to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China